CLINICAL TRIAL: NCT03573193
Title: Radiographic Bone Changes Following Socket Preservation in Mandibular Molars Using Deproteinized Bovine Bone Mineral Versus Using Beta Tri Calcium Phosphate
Brief Title: Radiographic Changes Following Socket Preservation in Molars Using Bovine Bone Versus Using Beta Tri ca.ph
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, wahid yehia al azizy al hussiney, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: socket preservation
Record Dates: First submitted 2018-06-13; First posted 2018-06-29 (Actual); Last update posted 2018-06-29 (Actual); Status verified 2018-06

CONDITIONS: Socket Preservation
Keywords: xenograft bone; synthetic bone substitutes

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial.
  • Unicenter, single blinded, with equal randomization, active controlled, parallel group study
Who Masked: Participant
Masking Description: Blinded participants
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group: (Active Comparator): ridge preservation alveolar ridge socket preserved using alloplastic material beta tri calcium phosphate type
  Interventions: Other: ridge preservation
- control group (Other): ridge preservation (alveolar ridge socket preserved using xenograft material Bio-oss type
  Interventions: Other: ridge preservation

INTERVENTIONS:
Other: ridge preservation — Intra operative procedures (for both groups) ridge preservation
  * Local anesthesia will be given to the patient.
  * Scrubbing and draping of the patient will be carried out in a standard fashion for intra oral procedures.
  * A crestal incision was made, and a mucoperiosteal flap was elevated. Implant osteotomies were prepared according to the recommendations and desired dimensions of implants.
  * In study group: tooth extraction with ridge preservation using deproteinized bovine bone mineral Bio-Oss
  * In the comparators group: tooth extraction with ridge preservation using an alloplastic ceramic material beta tricalcium phosphate (TCP).

SUMMARY:
Inadequate ridge width to allow implant placement, it noted that when extraction takes place and ridge preservation is not utilized the site of extraction could lose 40% to 60% of bone height and width within 2 to 3 years and subsequent loss of 0.25% to 0.5% annually. it reported as much as 4 mm loss of ridge width in extraction alone sites within 6 months. Using an atraumatic tooth extraction technique preserves osseous walls thereby improving the chances of osseous graft success.

The goal of ridge preservation is minimizing bone loss to preserve the maximum final, healed ridge dimensions.

Socket preservation is done using a hard tissue graft like xenograft bone or synthetic bone substitutes and prevent hazard of surgical intervention which needed during implant loading due to bone resorption.

DETAILED DESCRIPTION:
Good assessment whether a particular graft is more beneficial than others which can be improve the extraction site healing.

Good assessment if grafting has any beneficial or detrimental effects on post-operative sequelae post extraction.

Extraction is indicated when a tooth cannot be restored or maintained in suitable conditions for long-term health, function, and/or esthetics. Loss of a tooth has a direct effect on life quality by impairing the ability to masticate, speak, and, in some instances, socialize, after tooth extraction an average alveolar bone loss of 1.5-2 mm (vertical) and 40%-50% (horizontal) occurs within 6 months, alveolar dimensional changes occur during the first 3 months. If no treatment to restore the dentition is provided, then continued bone loss occurs and up to 40%-60% of ridge volume is lost in first 3 years . And the absence of a tooth in its alveolus enhances a cascade of biological events that typically result in significant local anatomic changes..

Studies have demonstrated that loss of alveolar ridge Post extraction is an irreversible process result in both horizontal and vertical reduction. Atrophy of alveolar ridge may have a significant effect on tooth replacement therapy, especially when implant restorations are planned.

Therefore, alveolar ridge preservation has become a key component of contemporary clinical dentistry.

Past therapy attempts to prevent resorption of alveolar ridge were performed by root retention, with the primary goal of maximizing the stability of removable prostheses. In spite of that, root retention is not always practical because of fracture, caries, and/or strategic reasons.

Alveolar ridge preservation via "socket grafting" started in the mid-1980s as a therapeutic alternative to root submergence. Its use was rationalized on the opinion that "filling" the space left by the extracted tooth with a biomaterial would simulate a "root retention effect" conducive to bone preservation, which would subsequently facilitate placement of implant by reducing the need of additional grafting procedures. This approach gained popularity over the years because of its conceptual attractiveness and simple technical procedures.

Over the past twenty years, multiple studies evaluating the efficacy of different socket-filling access have been conducted. In these studies, many of biomaterials have been employed, including autologous bone, bone substitutes (allografts, xenografts, and alloplasts), bioactive agents, and autologous blood-derived products.

Use of a grafting material with or without a membrane (alveolar ridge preservation) give additional support for stabilization of blood clot and space maintenance, bone loss is reduced from 69% to 25% or less. Objective of alveolar ridge preservation reduces bone loss, reduce the need for additional bone, and provide soft tissue support. And sinus augmentation procedures . finally providing for easier implant placement and a higher potential of achieving an esthetic restorative outcome.

Ridge preservation procedures are indicated when buccal plate thickness less than 1.5-2mm (most anterior and esthetic zones), damage or loss of one or more socket walls, maintaining bone volume is crucial to minimize the risk to adjacent anatomical structures, patients where many teeth are being extracted and preservation of bone is important for further restoration, and patients with high esthetic demands such as a high lip line and thin biotype, which are more prone to tissue loss.

Xenogenic Bone Grafts (Xenografts): Xenografts are derived from other species; Grafts are harvested from animals, mainly cows. That is why this is processed to make it totally biocompatible and sterile.

Advantages of xenografts:

- Only one simple procedure is needed as the bone is not being harvested from the patient in dangerous surgical procedures and it will encourage Natural bone growth.

Disadvantage of xenografts:

Is the minimal risk of bovine sponge form encephalopathy due to the fact that all organic components of the bone are extracted? The most widely used xenograft bone is deproteinized bovine bone mineral. Xenograft bone has similar properties to human cancellous bone, in its crystalline content and its macrostructure; it also has similar physical properties to the human bone This is a purely mineral graft and is osteoconductive but also some resorption will happen, so its use also has limitation. When used in a particulate form it is mixed with the patient's blood and packed into the defect.

They are materials with their organic components totally removed, With their removal, concern about immunological reactions becomes nonexistent, The remaining inorganic structure provides a natural architectural matrix as well as an excellent source of calcium The inorganic material also maintains the physical dimension of the augmentation during the remodeling phases.

choice of comparators: Alloplasts are synthetic bone substitutes. They are made of inorganic biocompatible materials including synthetic hydroxyapatite, tricalcium phosphate, bioactive glass, and calcium carbonate. Whether synthetic hydroxyapatite is resorbable or nonresorbable depends on the temperature at which it is prepared.

High-temperature preparation of hydroxyapatite results in a nonresorbable, dense material, nonporous, which is used as filler. Tricalcium phosphate acts as filler and is partially resorbable. Calcium carbonate, which is derived from coral, is biocompatible and resorbable so that it acts as filler, which eventually may be replaced by new bone. Bioactive glass is a silicone-based, osteoconductive material that bonds to bone through the formation of carbonated hydroxyapatite.

The advantage of alloplasts is that they have no potential for disease transmission.

Among the most promising is the tricalcium phosphate , an alloplastic ceramic material studied and used extensively in the past decade. It is considered to be bioactive (by means of inducing specific biologic reactions) and (not stimulating inflammatory or foreign-body giant cell activity) biocompatible.

This is mainly because tricalcium phosphate is composed of Ca and P ions, which are the most commonly found elements in bone. However, tricalcium phosphate cements have a slower resorption rate than bone and are usually too dense to allow bone tissue to grow into the defect in a limited period of time.

By adding a faster resorbing material, pores may be created, ensuring new bone tissue growing into the defect.

Tricalcium phosphate as a bone graft substitute has been evaluated at length in previous studies. It binds to bone by means of mechanical anchorage with no formation of intermediate apatite layer. Bioresorption of tricalcium phosphate granules occurs due to chemical dissolution in biological fluids and cellular degradation.

Solubilization is induced by mesenchymal cells, which are also actively involved in the degradation process.

the capability of osteoplastic cells, fibroblasts, and osteoclasts to degrade TCP ceramic material. Monocyte/macrophage participation is well documented in vivo as well as in vitro.

It seems that the more soluble a CaP ceramic, the more rapidly it is resorbed by osteoclasts. However, the increased number of released calcium ions may, on one hand, inhibit osteoclasts' activity, while on the other hand, it provides a good environment for osteogenesis. Therefore, it seems that Tricalcium phosphate resorption is performed at a rather unpredictable rate that does not always correspond to the new bone formation rate. This behavior is evident in the conflicting results of many studies on the bioresorption of TCP.

The βeta- phase isomer of Tricalcium phosphate (β -Tricalcium phosphate ), however, is characterized by homogenous microporosity, physiologic pH, increased solubility, and a more predictable resorption rate that look alike the new bone remodeling rate. Composition or impurities Variations may affect solubility, whereas the pure phase seems to be resorbed in 5 to 6 months.

It should be noted that a faster resorbable material might allow soft-tissue cells to prematurely intrude into the defect, while slowly resorbable or nonresorbable materials that remain for a long time may inhibit new bone deposition.

ELIGIBILITY:
Inclusion Criteria:

* Good oral hygiene.
* Age from 25-60 years
* Both sexes
* Sufficient bone volume
* Presence of non-restorable mandibular molars.

Exclusion Criteria

* Extreme bone atrophy.
* Patients who have systemic disorders that might interfere with bone metabolism.
* Pregnant patients.
* Bad oral hygiene.
* Patients with bone diseases.
* Patient with limited mouth opening

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-07 (Estimated); Primary Completion 2018-11 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Prevent post extraction ridge volume loss and decrease bone resorption detected by CBCT to prepare for success implant loading | base lline
  socket preservation is minimizing bone loss to preserve the maximum final, healed ridge dimensions

CONTACTS AND LOCATIONS:
Overall Officials: AMR A al azim, professor, Study Director — Cairo University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gerritsen AE, Allen PF, Witter DJ, Bronkhorst EM, Creugers NH. Tooth loss and oral health-related quality of life: a systematic review and meta-analysis. Health Qual Life Outcomes. 2010 Nov 5;8:126. doi: 10.1186/1477-7525-8-126. PMID 21050499
- [Result] Schropp L, Wenzel A, Kostopoulos L, Karring T. Bone healing and soft tissue contour changes following single-tooth extraction: a clinical and radiographic 12-month prospective study. Int J Periodontics Restorative Dent. 2003 Aug;23(4):313-23. PMID 12956475
- [Result] Van der Weijden F, Dell'Acqua F, Slot DE. Alveolar bone dimensional changes of post-extraction sockets in humans: a systematic review. J Clin Periodontol. 2009 Dec;36(12):1048-58. doi: 10.1111/j.1600-051X.2009.01482.x. PMID 19929956
- [Result] Seibert JS, Salama H. Alveolar ridge preservation and reconstruction. Periodontol 2000. 1996 Jun;11:69-84. doi: 10.1111/j.1600-0757.1996.tb00185.x. No abstract available. PMID 9567959
- [Result] Osburn RC. Preservation of the alveolar ridge: a simplified technique for retaining teeth beneath removable appliances. J Indiana State Dent Assoc. 1974 Jan-Feb;53(1):8-11. No abstract available. PMID 4523604
- [Result] Artzi Z, Nemcovsky CE. The application of deproteinized bovine bone mineral for ridge preservation prior to implantation. Clinical and histological observations in a case report. J Periodontol. 1998 Sep;69(9):1062-7. doi: 10.1902/jop.1998.69.9.1062. PMID 9776036
- [Result] Christensen GJ. Ridge preservation: why not? J Am Dent Assoc. 1996 May;127(5):669-70. doi: 10.14219/jada.archive.1996.0279. PMID 8642146
- [Result] Darby I, Chen ST, Buser D. Ridge preservation techniques for implant therapy. Int J Oral Maxillofac Implants. 2009;24 Suppl:260-71. PMID 19885449
- [Result] Tallgren A. The continuing reduction of the residual alveolar ridges in complete denture wearers: a mixed-longitudinal study covering 25 years. J Prosthet Dent. 1972 Feb;27(2):120-32. doi: 10.1016/0022-3913(72)90188-6. No abstract available. PMID 4500507
- [Result] Hammerle CH, Araujo MG, Simion M; Osteology Consensus Group 2011. Evidence-based knowledge on the biology and treatment of extraction sockets. Clin Oral Implants Res. 2012 Feb;23 Suppl 5:80-2. doi: 10.1111/j.1600-0501.2011.02370.x. PMID 22211307
- [Result] De Buitrago JG, Avila-Ortiz G, Elangovan S. Quality assessment of systematic reviews on alveolar ridge preservation. J Am Dent Assoc. 2013 Dec;144(12):1349-57. doi: 10.14219/jada.archive.2013.0070. PMID 24282264
- [Result] Omran M, Min S, Abdelhamid A, Liu Y, Zadeh HH. Alveolar ridge dimensional changes following ridge preservation procedure: part-2 - CBCT 3D analysis in non-human primate model. Clin Oral Implants Res. 2016 Jul;27(7):859-66. doi: 10.1111/clr.12701. Epub 2015 Oct 25. PMID 26498407
- [Result] Barone A, Orlando B, Cingano L, Marconcini S, Derchi G, Covani U. A randomized clinical trial to evaluate and compare implants placed in augmented versus non-augmented extraction sockets: 3-year results. J Periodontol. 2012 Jul;83(7):836-46. doi: 10.1902/jop.2011.110205. Epub 2011 Dec 5. PMID 22141358
- [Result] Rasperini G, Canullo L, Dellavia C, Pellegrini G, Simion M. Socket grafting in the posterior maxilla reduces the need for sinus augmentation. Int J Periodontics Restorative Dent. 2010 Jun;30(3):265-73. PMID 20386783
- [Result] Darby I, Chen S, De Poi R. Ridge preservation: what is it and when should it be considered. Aust Dent J. 2008 Mar;53(1):11-21. doi: 10.1111/j.1834-7819.2007.00008.x. PMID 18304236
- [Result] Nazirkar G, Singh S, Dole V, Nikam A. Effortless effort in bone regeneration: a review. J Int Oral Health. 2014 Jun;6(3):120-4. Epub 2014 Jun 26. PMID 25083047
- [Result] Zaner DJ, Yukna RA. Particle size of periodontal bone grafting materials. J Periodontol. 1984 Jul;55(7):406-9. doi: 10.1902/jop.1984.55.7.406. PMID 6086869
- [Result] Callan DP, Rohrer MD. Use of bovine-derived hydroxyapatite in the treatment of edentulous ridge defects: a human clinical and histologic case report. J Periodontol. 1993 Jun;64(6):575-82. doi: 10.1902/jop.1993.64.6.575. PMID 8393110
- [Result] Esposito M, Grusovin MG, Felice P, Karatzopoulos G, Worthington HV, Coulthard P. Interventions for replacing missing teeth: horizontal and vertical bone augmentation techniques for dental implant treatment. Cochrane Database Syst Rev. 2009 Oct 7;2009(4):CD003607. doi: 10.1002/14651858.CD003607.pub4. PMID 19821311
- [Result] Cameron HU, Macnab I, Pilliar RM. Evaluation of biodegradable ceramic. J Biomed Mater Res. 1977 Mar;11(2):179-86. doi: 10.1002/jbm.820110204. PMID 853042
- [Result] Jarcho M. Biomaterial aspects of calcium phosphates. Properties and applications. Dent Clin North Am. 1986 Jan;30(1):25-47. PMID 3514291
- [Result] LeGeros RZ. Properties of osteoconductive biomaterials: calcium phosphates. Clin Orthop Relat Res. 2002 Feb;(395):81-98. doi: 10.1097/00003086-200202000-00009. PMID 11937868
- [Result] Nilsson M, Fernandez E, Sarda S, Lidgren L, Planell JA. Characterization of a novel calcium phosphate/sulphate bone cement. J Biomed Mater Res. 2002 Sep 15;61(4):600-7. doi: 10.1002/jbm.10268. PMID 12115450
- [Result] Artzi Z, Weinreb M, Givol N, Rohrer MD, Nemcovsky CE, Prasad HS, Tal H. Biomaterial resorption rate and healing site morphology of inorganic bovine bone and beta-tricalcium phosphate in the canine: a 24-month longitudinal histologic study and morphometric analysis. Int J Oral Maxillofac Implants. 2004 May-Jun;19(3):357-68. PMID 15214219
- [Result] Kotani S, Fujita Y, Kitsugi T, Nakamura T, Yamamuro T, Ohtsuki C, Kokubo T. Bone bonding mechanism of beta-tricalcium phosphate. J Biomed Mater Res. 1991 Oct;25(10):1303-15. doi: 10.1002/jbm.820251010. PMID 1812121
- [Result] Evans RW, Cheung HS, McCarty DJ. Cultured human monocytes and fibroblasts solubilize calcium phosphate crystals. Calcif Tissue Int. 1984 Dec;36(6):645-50. doi: 10.1007/BF02405384. PMID 6442200
- [Result] Owens JL, Cheung HS, McCarty DJ. Endocytosis precedes dissolution of basic calcium phosphate crystals by murine macrophages. Calcif Tissue Int. 1986 Mar;38(3):170-4. doi: 10.1007/BF02556877. PMID 3085894
- [Result] Gregoire M, Orly I, Menanteau J. The influence of calcium phosphate biomaterials on human bone cell activities. An in vitro approach. J Biomed Mater Res. 1990 Feb;24(2):165-77. doi: 10.1002/jbm.820240204. PMID 2329113
- [Result] Gaasbeek RD, Toonen HG, van Heerwaarden RJ, Buma P. Mechanism of bone incorporation of beta-TCP bone substitute in open wedge tibial osteotomy in patients. Biomaterials. 2005 Nov;26(33):6713-9. doi: 10.1016/j.biomaterials.2005.04.056. PMID 15950278
- [Result] Fujita R, Yokoyama A, Nodasaka Y, Kohgo T, Kawasaki T. Ultrastructure of ceramic-bone interface using hydroxyapatite and beta-tricalcium phosphate ceramics and replacement mechanism of beta-tricalcium phosphate in bone. Tissue Cell. 2003 Dec;35(6):427-40. doi: 10.1016/s0040-8166(03)00067-3. PMID 14580356
- [Result] Bowers GM, Vargo JW, Levy B, Emerson JR, Bergquist JJ. Histologic observations following the placement of tricalcium phosphate implants in human intrabony defects. J Periodontol. 1986 May;57(5):286-7. doi: 10.1902/jop.1986.57.5.286. PMID 3457941
- [Result] Rey C. Calcium phosphate biomaterials and bone mineral. Differences in composition, structures and properties. Biomaterials. 1990 Jul;11:13-5. PMID 2397252
- [Result] Trisi P, Rao W, Rebaudi A, Fiore P. Histologic effect of pure-phase beta-tricalcium phosphate on bone regeneration in human artificial jawbone defects. Int J Periodontics Restorative Dent. 2003 Feb;23(1):69-77. PMID 12617370